CLINICAL TRIAL: NCT03533699
Title: A Comparison Between the Effect of Oxytocin Only and Oxytocin Plus Propranolol on Induction of Labor in Term Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: propranolol, labor induction
Record Dates: First submitted 2018-04-23; First posted 2018-05-23 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Propranolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Intervention Model Description: In the first group (Propranolol plus Oxytocin), a capsule consisting of 20 mg Propranolol will be administered and in the second group (Oxytocin plus placebo), a similar capsule as a placebo will be administrated orally by researcher before beginning of induction of labour.
  Induction will be initiated at a dose of 2 mIu/min and it will be increased 2 mIu / minute every 15 minutes until good contractions are obtained (3 forceful contractions within 10 minutes) or to a maximum dose of 30 mIu/min; then, it will be continued at this rate for 8 hours. If patients enter the active phase of labour (cervical dilatation = 3-4 cm), induction will be continued until delivery. If no response to induction of labour, a caesarean section will be performed.
Who Masked: Participant, Investigator
Masking Description: Then Patients will be randomly assigned to two groups using sealed, sequentially distributed envelopes to which the letters A and B will be allocated. The letter A will be assigned to the propranolol group and the letters B to the oxytocin group. The envelopes, will be opened by the investigator, and according to the letters, the group of patients will be determined. The first vaginal examination will be performed by the investigator, and then the induction will be initiated by the same researcher. Continuation of induction and the control of patients will be monitored by a coworker who knew nothing about the method of initiation of induction, neither did the patients (double blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol (Active Comparator): 101 women with uncomplicated term pregnancy who will be admitted to the Ain Shams University Maternity hospital and will receive syntocinon intravenous infusion for induction or augmentation of labour.
  Interventions: Drug: Propranolol
- placebo (Placebo Comparator): 101 women with uncomplicated term pregnancy who will be admitted to the Ain Shams University Maternity hospital and will receive syntocinon intravenous infusion for induction or augmentation of labour.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Propranolol
  Other Names: beta blocker; indral
  Arms: Propranolol
Drug: Placebo Oral Tablet — oral tablets with no active drug
  Arms: placebo

SUMMARY:
The present study is conducted to compare the effect of Oral Propranolol and Oxytocin, versus Oxytocin only on induction of labor in term pregnancy.

DETAILED DESCRIPTION:
After receiving approval from the Hospital Ethics Committee, women with uncomplicated term pregnancy who will be admitted to the Ainshams maternity hospital will be recruited in this study.

Inclusion criteria:

1. Gestational age of 38-41 weeks of pregnancy (according to a reliable last menstrual period (LMP) and sonography of first trimester)
2. Nulliparity,
3. Singleton pregnancy.
4. Cephalic presentation.
5. Intact membranes.
6. Bishop Score 5 or more.

Exclusive criteria:

1. Pelvic contraction,
2. Previous surgical operation on the uterus,
3. Signs of fetal distress,
4. Placenta previa
5. Suspicious macrosomia,
6. Polyhydramnios,
7. Hydrocephalus of fetus
8. History of any known cardiac, pulmonary or metabolic disorder of mother, or maternal drug use.

Sample size calculation:

Assuming an effect size regarding interval until good contractions of 0.6(Ashraf DM et al., 2013), a sample size of 101 in each group would be enough to elucidate such effect if true, at 0.05 alpha error and 0.95 power of the test. Sample size could be inflated by 10% for dropouts so the total would be 112 in each group Sample size was calculated using sample size table calculation in designing clinical research appendix 6A (Hulley, S.B. et al., 2013)

Intervention to be done:

After taking informed consent, all pregnant ladies recruited in the study will undergo complete clinical examination and detailed medical history will be obtained along with necessary lab investigations and ultrasound findings. Each patient will have a case record form in which the following data will be recorded:

• History: Personal (age, duration of marriage), present (any current medical or surgical diseases and any current medication), obstetric history (Gestational age, obstetric complications) and past history (cardiac, pulmonary or metabolic diseases).

* Clinical examination:

  1. General examination: assessment of vital data, cardiac and chest auscultation to exclude contraindications for drug administration.
  2. Abdominal examination: assessment of fundal level and contractions.
  3. PV examination: assessment of Bishop score, membranes status and fetal presentation.
* Investigations:

  1. Routine investigations will be done e.g., complete blood count and blood grouping.
  2. Pelvi-abdominal U/S (Confirm fetal life, placental location, fetus parameters, amniotic fluid index and expected fetal weight).
* Confirmation of gestational age before 20 weeks' gestation (regular menstrual history with known last menstrual period and/or ultrasound confirmation of gestational age by means of crown rump length measurement in 1st trimester).
* Assessment of uterine contractions and PV examination (cervical dilation and effacement, station of fetal head, fetal presentation, membranes status) are done and recorded and bishop score will be measured.
* CTG will be done for all pregnant ladies included in the study.
* Randomization:

Then Patients will be randomly assigned to two groups using sealed, sequentially distributed envelopes to which the letters A and B will be allocated. The letter A will be assigned to the propranolol group and the letters B to the oxytocin group. The envelopes, will be opened by the investigator, and according to the letters, the group of patients will be determined. The first vaginal examination will be performed by the investigator, and then the induction will be initiated by the same researcher. Continuation of induction and the control of patients will be monitored by a coworker who knew nothing about the method of initiation of induction, neither did the patients (double blind)

In the first group (Propranolol plus Oxytocin), a capsule consisting of 20 mg Propranolol will be administered and in the second group (Oxytocin plus placebo), a similar capsule as a placebo will be administrated orally by researcher before beginning of induction of labour.

Induction will be initiated at a dose of 2 mIu/min and it will be increased 2 mIu / minute every 15 minutes until good contractions are obtained (3 forceful contractions within 10 minutes) or to a maximum dose of 30 mIu/min; then, it will be continued at this rate for 8 hours. If patients enter the active phase of labour (cervical dilatation = 3-4 cm), induction will be continued until delivery. If no response to induction of labour, a caesarean section will be performed.

Blood pressures and heart rate of the parturients and fetal heart rates will be monitored every 15 minutes. The participants' characteristics, age, primary Bishop score, gestational age, the number of deliveries on the first day of induction and caesarean sections, timing of the beginning good contractions after induction, duration of latent phase (interval between the beginnings of good contractions until cervical dilatations of 3-4 cm will be obtained), type of delivery and Apgar scores of minutes 1 and 5, need of admissions to NICU and neonatal weights will be recorded and compared in the two groups. The participants will be followed up until delivery.

The partogram will be used to monitor the fetal heart rate, membranes status, cervical dilation and effacement, station of the fetus and uterine contractions (rate and strength).

After delivery mothers will be encouraged to establish skin to skin contact and breast feeding as soon as possible after birth. Babies will be encouraged to feed on demand but the interval between feeds will be no longer than 3 hours Samples for measuring blood glucose level for the newborn will be taken 1 hour after birth regardless of feeds, then before feeds 3-4 hourly in the first 24 hours. Measurements will be discontinued if there are 3 normal blood glucose concentration measurements and no clinical concerns about feeding.

Also fetal heart rate will be measured every 4 hours for 24 hours after delivery

Safety considerations:

If the parturient has hyperstimulation of contractions (in a situation with more than 5 contractions/10 mins, duration of contractions <90 secs, interval of contraction less than 2 min or fetal distress) the augmentation will be stopped and the parturient is kept in left lateral position and given oxygen, and intravenous dextrose.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age of 38-41 weeks of pregnancy (according to a reliable last menstrual period (LMP) and sonography of first trimester)
2. Nulliparity,
3. Singleton pregnancy.
4. Cephalic presentation.
5. Intact membranes.
6. Bishop Score 5 or more.

Exclusion Criteria:

1. Pelvic contraction,
2. Previous surgical operation on the uterus,
3. Signs of fetal distress,
4. Placenta previa
5. Suspicious macrosomia,
6. Polyhydramnios,
7. Hydrocephalus of fetus
8. History of any known cardiac, pulmonary or metabolic disorder of mother, or maternal drug use.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 202 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Time from active phase to delivery in minutes | 16 hours
  Time from active phase to delivery in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No